CLINICAL TRIAL: NCT02940847
Title: The Effectiveness of Ultrasound-guided Technique Compared to Blind Technique in Medial Brachial Cutaneous Nerve Block and Intercostobrachial Nerve Block, in the Axilla
Brief Title: Ultrasound-guided Versus Blind Technique in Medial Brachial Cutaneous Nerve and Intercostobrachial Nerve Blocks
Acronym: ECHO_NCMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-A01296-45
Record Dates: First submitted 2016-10-16; First posted 2016-10-21 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Upper Limb Surgery
Keywords: ultrasound-guided technique; blind technique; medial brachial cutaneous nerve block; intercostobrachial nerve block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- blind technique (Active Comparator): Investigators will perform a medial brachial cutaneous nerve block and an intercostobrachial nerve block with either a blind technique or an ultrasound-guided technique to estimate the effectiveness of each technique. The blind technique consists in performing a subcutaneous injection of the local anesthetic at the root of the arm, in the anterior-posterior direction.
  Interventions: Procedure: medial brachial cutaneous nerve block and intercostobrachial nerve block with blind technique
- ultrasound-guided technique (Active Comparator): Investigators will perform a medial brachial cutaneous nerve block and an intercostobrachial nerve block with either a blind technique or an ultrasound-guided technique to estimate the effectiveness of each technique. In the ultrasound-guided technique, ultrasounds are used to visualize the anatomical variations, the good position of the needle and the good local anesthetic diffusion.
  Interventions: Procedure: medial brachial cutaneous nerve block and intercostobrachial nerve block with ultrasound-guided technique

INTERVENTIONS:
Procedure: medial brachial cutaneous nerve block and intercostobrachial nerve block with blind technique — It consists in performing a subcutaneous injection of the local anesthetic at the root of the arm, in the anterior-posterior direction.
  Arms: blind technique
Procedure: medial brachial cutaneous nerve block and intercostobrachial nerve block with ultrasound-guided technique — Ultrasounds are used to visualize the anatomical variations, the good position of the needle and the good local anesthetic diffusion.
  Arms: ultrasound-guided technique

SUMMARY:
The axillary brachial plexus block is a technique of locoregional anesthesia indicated in the distal upper limb surgery : hand, forearm, the lower third of the arm including the elbow. The anesthesia of the posterior and the medial side of the arm requires a selective block of the medial brachial cutaneous nerve and the intercostobrachial nerve, for example to improve the tolerance of the inflatable tourniquet used by the surgeons. There are two techniques to achieve this block : the blind technique (without ultrasound) and the ultrasound-guided technique. At the moment, there are no studies which compare these two techniques. So, the purpose of this study is to determine the effectiveness of ultrasound-guided technique compared to blind technique in medial brachial cutaneous nerve block and intercostobrachial nerve block, in the axilla.

DETAILED DESCRIPTION:
For purposes of this single-blind monocentric study, 84 patients are randomized into two groups (42 patients for each), upon enrolment into the study.

In the first group, the blind technique is used to perform the medial brachial cutaneous nerve block and the intercostobrachial nerve block : it consists in performing a subcutaneous injection of the local anesthetic at the root of the arm, in the anterior-posterior direction.

In the second group, the ultrasound-guided technique is used to perform the medial brachial cutaneous nerve block and the intercostobrachial nerve block : ultrasounds are used to visualize the anatomical variations, the good position of the needle and the good local anesthetic diffusion.

The aim is to evaluate the effectiveness of ultrasound-guided technique compared to blind technique in medial brachial cutaneous nerve block and intercosto-brachial nerve block, in the axilla

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years
* Surgery of the distal upper limb : hand, forearm, lower third of the arm ,including the elbow
* Urgent or planned surgery
* Locoregional anesthesia : axillary brachial plexus block, completed by a medial brachial cutaneous nerve block and an intercostobrachial nerve block
* Local anesthetic used : mepivacaine 10mg/ml
* In the absence of patient objections

Exclusion Criteria:

* Pregnancy
* Adults under guardianship
* Locoregional anesthesia contraindications
* Local anesthetic used : ropivacaine 0,75%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-11-13 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with complete anesthesia in the lower half of the medial cutaneous area of the arm, at time 20 minutes | at time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block
  At time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block, a light touch sensitivity test is performed
Number of participants with complete anesthesia in the upper half of the medial cutaneous area of the arm, at time 20 minutes | at time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block
  At time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block, a light touch sensitivity test is performed
Number of participants with complete anesthesia in the lower half of the posterior cutaneous area of the arm, at time 20 minutes | at time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block
  At time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block, a light touch sensitivity test is performed
Number of participants with complete anesthesia in the upper half of the posterior cutaneous area of the arm, at time 20 minutes | at time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block
  At time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block, a light touch sensitivity test is performed
Number of participants with complete anesthesia of the arm at time 20 minutes | at time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block
  At time 20 minutes after the achievement of medial brachial cutaneous nerve block and intercostobrachial nerve block, a light touch sensitivity test is performed

SECONDARY OUTCOMES:
Number of participants with complete anesthesia, with reduced sensitivity and with absence of anesthesia at times 5, 10, 15, 20 minutes (except primary outcome) in the areas of the medial brachial cutaneous nerve and the intercostobrachial nerve | at times 5, 10, 15, 20 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
Number of patients with comfortable feeling, with unpleasant sensations and with pains during surgery, in the areas of the medial brachial cutaneous nerve and the intercostobrachial nerve (questionnaire completed by the anesthesist) | 3 hours after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
The total volume (mL) of local anesthetic used for the medial brachial cutaneous nerve block and the intercostobrachial nerve block | 5 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
Number of participants (of the ultrasound-guided group) with good ultrasound view of theses nerves before and after the injection of the local anesthetic | 5 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
Number of participants (of the ultrasound-guided group) with : bad ultrasound view of theses nerves before the injection and good ultrasound view of theses nerves after the injection of the local anesthetic | 5 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
Number of participants (of the ultrasound-guided group) with bad ultrasound view of theses nerves before and after the injection of the local anesthetic. | 5 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Hervé BOUAZIZ, Professor, Study Director — CHU NANCY
Locations (1):
- Chru Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magazzeni P, Jochum D, Iohom G, Mekler G, Albuisson E, Bouaziz H. Ultrasound-Guided Selective Versus Conventional Block of the Medial Brachial Cutaneous and the Intercostobrachial Nerves: A Randomized Clinical Trial. Reg Anesth Pain Med. 2018 Nov;43(8):832-837. doi: 10.1097/AAP.0000000000000823. PMID 29905631